CLINICAL TRIAL: NCT04068766
Title: Efficacy of Paracervical Block in Laparoscopic Myomectomy: a Randomized Controlled Trial (PALM)
Acronym: PALM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KBSMC 2019-08-024
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Uterine Fibroid
MeSH Terms: conditions — Leiomyoma | interventions — Anesthesia, Obstetrical; Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paracervical block with 5% bupivacaine (Experimental): The paracervical injection with 10 mL of 0.5% bupivacaine plus 1:200,000 epinephrine was administrated by the second assistant surgeon into the cervicovaginal junction at 3 and 9 o'clock with a depth of 1 cm after intubation but before fixation of uterine manipulator onto the cervix.
  Interventions: Device: Paracervical block; Drug: 5% bupivacaine
- Paracervical block with normal saline (Placebo Comparator): ck with a depth of 1 cm after intubation but before fixation of uterine manipulator onto the cervix.
  Interventions: Device: Paracervical block; Drug: Normal saline

INTERVENTIONS:
Device: Paracervical block — The paracervical injection with 10 mL of 0.5% bupivacaine plus 1:200,000 epinephrine or normal saline was administrated by the second assistant surgeon into the cervicovaginal junction at 3 and 9 o'clock with a depth of 1 cm after intubation but before fixation of uterine manipulator onto the cervix.
  Other Names: Experimental arm; Control arm
Drug: 5% bupivacaine — The paracervical injection with 10 mL of 0.5% bupivacaine plus 1:200,000 epinephrine was administrated by the second assistant surgeon into the cervicovaginal junction at 3 and 9 o'clock with a depth of 1 cm after intubation but before fixation of uterine manipulator onto the cervix.
  Other Names: Experimental arm
  Arms: Paracervical block with 5% bupivacaine
Drug: Normal saline — The paracervical injection with 10 mL of normal saline was administrated by the second assistant surgeon into the cervicovaginal junction at 3 and 9 o'clock with a depth of 1 cm after intubation but before fixation of uterine manipulator onto the cervix.
  Other Names: Control arm
  Arms: Paracervical block with normal saline

SUMMARY:
It remains controversial whether paracervical block should be performed as a powerful strategy for pain relief in laparoscopic myomectomy (LM), because convincing conclusions are difficult to draw because of the heterogeneous and contradictory nature of the literature. Therefore, the aim of this study was to evaluate the efficacy of paracervical blocks using with 0.5% bupivacaine prior to LM for benign gynecologic conditions on postoperative pain relief.

DETAILED DESCRIPTION:
However, no study investigating the efficacy of paracervical block in laparoscopic myomectomy on postoperative pain was conducted, to date. Therefore, the goal of this study is to evaluate whether patients who receive a paracervical block of 5% bupivacaine with epinephrine at the time of laparoscopic myomectomy would have lower postoperative pain, with less consumption of rescue analgesics than patients who receive a paracervical block of normal saline.

ELIGIBILITY:
Inclusion Criteria:

* Uterine myoma
* American Society of Anesthesiologists physical status (ASAPS) classification I-II
* The absence of pregnancy at the time of surgery.

Exclusion Criteria:

* history of cervical surgery such as conization or cerclage
* inability to perform the paracervical block due to anatomical abnormalities (i.e., very atrophic or small cervix)
* allergy to bupivacaine, planned concomitant surgical procedures involving extensive additional tissue manipulation such as pelvic lymph node dissection
* any concomitant surgery of pelvic floor repair (uterosacral ligament suspension or sacrocolpopexy) or vaginal procedure (anterior or posterior colporrhaphy or mid-urethral slings)
* previously taking opioids for chronic pain
* inability to accurately express their pain

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2019-08-23 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | at 6-hour after surgery
  The scale was presented as a 10-cm line with verbal descriptors ranging from "no pain" to "worst imaginable pain".

SECONDARY OUTCOMES:
Frequency of pills/injections requested | Within 24-hour after surgery
  Narcotic and non-narcotic use were measured by number of pills/injections requested within 24-hour after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, Principal Investigator — Kangbuk Samsung Hospital
Locations (2):
- South Korea (2):
  - Kangbuk Samsung Hospital, Seoul
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No